CLINICAL TRIAL: NCT02467582
Title: Adjuvant Aspirin Treatment in PIK3CA Mutated Colon Cancer Patients. A Randomized, Double-blinded, Placebo-controlled, Phase III Trial
Brief Title: Adjuvant Aspirin Treatment for Colon Cancer Patients
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Board decision in 2020 due to lack of financial funding.
Sponsor: Swiss Cancer Institute (Other)
Collaborators: European Organisation for Research and Treatment of Cancer - EORTC (Network); Central European Society for Anticancer Drug Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SAKK 41/13 - Aspirin; SNCTP000001339 (Registry Identifier: SNCTP); 2015-001482-57 (EudraCT Number)
Record Dates: First submitted 2015-06-05; First posted 2015-06-10 (Estimated); Results first posted 2025-05-16 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Colon Cancer
Keywords: Aspirin; colon cancer; stage II; stage III; PIK3CA; double-blind; placebo; Adjuvant Treatment
MeSH Terms: conditions — Colonic Neoplasms; Hereditary Sensory and Autonomic Neuropathies | interventions — Aspirin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aspirin 100 mg (Experimental): Asprin 100 mg daily for maximum 3 years standard chemo if indicated
  Interventions: Drug: Aspirin
- Placebo (Active Comparator): Placebo daily for maximum 3 years standard chemo if indicated
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Aspirin — Aspirin 100 mg daily
  Other Names: acetylsalicylic acid
  Arms: Aspirin 100 mg
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
Following complete resection of their primary tumor, potentially eligible stage II or stage III colon cancer patients will undergo central PIK3CA testing. Patients with somatic mutations will be 2:1 randomized to daily aspirin 100 mg versus placebo for a a maximum of 3 years or until disease recurrence, patient death or withdrawal of consent, whichever occurs first. Patients will be followed up for at least 3 years from the date of surgery.

The intake of aspirin or placebo is independent of adjuvant chemotherapy, and does not impact on the indication to give (or not to give) adjuvant chemotherapy.

DETAILED DESCRIPTION:
Colorectal cancer is the third most common malignancy for both women and men and is responsible for almost 10% of all cancer death. Despite complete removal of the tumor and use of adjuvant chemotherapy, up to 25% of patients with stage II colon cancer and up to 50% of patients with stage III disease will suffer from recurrences, which is associated with poor prognosis.

Several retrospective observations have documented a favorable effect of long-term intake of oral aspirin for the prevention of colorectal cancer in different clinical situations. Regular intake of aspirin after the diagnosis of colorectal cancer may also be associated with a lower risk of colorectal cancer-specific and overall mortality. Two recent publications in prestigious medical journals provided retrospective evidence that patients with PIK3CA-mutated colon cancer may derive a very substantial benefit from daily oral aspirin. Both analyses showed a roughly 85% reduction of the risk for tumor relapse compared to patients who did not take aspirin. However, a potential selection bias in these retrospective analyses cannot be excluded with certainty. These extremely interesting and intriguing findings must be confirmed in a randomized controlled trial to potentially change clinical practice.

The trial objective is to demonstrate a statistically significant and clinically relevant disease-free survival benefit in stage II and III PIK3CA mutated colon cancer patients taking daily adjuvant aspirin for 3 years.

Patients with resected colon cancer stage II or stage III bearing somatic mutations in exon 9 or 20 of PIK3CA will be 2:1 randomized to daily adjuvant aspirin 100 mg versus placebo for a maximum of 3 years or until disease recurrence, patient death or withdrawal of consent, whichever occurs first. Patients will be followed up for at least 3 years from the date of surgery. The intake of aspirin or placebo is independent of adjuvant chemotherapy, and does not impact on the indication to give (or not to give) adjuvant chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent according to ICH/GCP regulations before inclusion and prior to any trial-related investigations.
* Histologically confirmed diagnosis of adenocarcinoma of the colon.
* Stage II (pT3/T4 N0 cM0) or stage III (pTx pN+ cM0) colon cancer.
* Availability of cancer tissue for central molecular testing.
* Presence of predefined, activating PIK3CA mutation in exons 9 or 20 (centrally assessed).
* Complete resection of the primary tumor (R0) within 14 weeks maximum before registration.
* WHO performance status 0-2.
* Age between 18-80 years.
* Adequate hematological values: hemoglobin ≥ 80 g/L, platelets ≥ 50 x 109/L.
* Adequate hepatic function: total bilirubin ≤1.5xULN, AST ≤2.5xULN, ALT ≤2.5xULN, AP ≤2.5xULN.
* Calculated creatinine clearance > 30 mL/min, according to the formula of Cockcroft-Gault.
* Women with child-bearing potential are using effective contraception, are not pregnant or lactating and agree not to become pregnant during trial treatment. A negative pregnancy test before inclusion (within 7 days) into the trial is required for all women with child-bearing potential.

Exclusion Criteria:

* Previous or concomitant malignancy within 3 years of registration, except for adequately treated cervical carcinoma in situ or localized non-melanoma skin cancer.
* Multiple adenocarcinomas of the colon.
* Rectal cancer (defined as distance from anal verge to proximal/oral tumor edge ≤15 cm).
* Severe or uncontrolled cardiovascular disease (congestive heart failure NYHA III or IV, unstable angina pectoris, history of myocardial infarction) within three months prior to registration.
* Systemic rheumatic diseases or degenerative disorders affecting the musculoskeletal system with a relevant risk of requiring treatment with NSAIDs in the future.
* Comorbidities that require regular (i.e. more than 3x per month, any dose) intake of acetylsalicylic acid or other NSAIDs or COX-2 inhibitors.
* Clinically relevant upper gastro-intestinal bleeding within 12 months prior to registration.
* Presence of any bleeding disorder that is an absolute contraindication to the use of aspirin.
* General tendency to hypersensitivity and history of asthma triggered by salicylates or substances with a similar mechanism of action, and non-steroidal anti-inflammatory drugs in particular
* Any serious underlying medical condition, at the judgment of the investigator, which could impair the ability of the patient to participate in the trial (e.g. uncontrolled infection, active autoimmune disease, uncontrolled diabetes).
* Concurrent treatment with other experimental drugs or treatment in an interventional clinical trial within 30 days prior to trial entry. Concomitant use of adjuvant chemotherapy for stage III and high risk stage II colon cancer according to international treatment guidelines is allowed (chemotherapy regimens include intravenous 5-fluorouracil or oral capecitabine either alone or in combination with intravenous oxaliplatin).
* Psychiatric disorder precluding understanding of trial information, giving informed consent or interfering with compliance for oral drug intake.
* Any familial, sociological or geographical condition potentially hampering proper staging and compliance with the trial protocol.
* Known or suspected hypersensitivity to any component of the trial drug or any agent given in association with this trial.
* Known galactose-1-phosphate uridyl transferase deficiency, UDP galactose 4 epimerase deficiency, galactokinase deficiency, orFanconi-Bickel syndrome, congenital lactase deficiency,or glucose-galactose malabsorption (due to the lactose-containing placebo).
* Any concomitant drugs contraindicated for use with the trial drug according to the approved product information.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1040 (Actual)
Dates: Start 2016-06-09 (Actual); Primary Completion 2023-09-14 (Actual); Study Completion 2023-09-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ulrich Güller, Prof, Study Chair — Spital STS AG Thun
Locations (60):
- Belgium (6):
  - Hopital Universitaire Brugmann, Brussels
  - Universitair Ziekenhuis Brussel, Brussels
  - Hôpital de Jolimont, Haine-Saint-Paul
  - CHC - Clinique Saint-Joseph, Liège
  - Az Damiaan, Ostend
  - AZ Turnhout - Campus Sint-Elisabeth, Turnhout
- Germany (23):
  - Spandau Vivantes Klinikum, Berlin
  - Fürst-Stirum-Klinik Bruchsal, Bruchsal
  - pioh KÖLN, Cologne
  - Universitätsklinikum Dresden, Dresden
  - Kliniken Essen Mitte, Essen
  - pioh Frechen, Frechen
  - Praxis und Tagesklinik - Medizinische Management GmbH, Friedrichshafen
  - Überörtliche Gemeinschaftspraxis - Schwerpunkt Haematologie, internistische Onkologie & Palliativmedizin, Hamburg
  - Universitätsklinikum Hamburg-Eppendorf, Hamburg
  - Medizinische Hochschule Hannover, Hanover
  - Onkologische Schwerpunktpraxis Heidelberg, Heidelberg
  - Onkologie UnterEms, Leer
  - Klinikum Ludwigsburg, Ludwigsburg
  - Universitätsmedizin Mannheim, Mannheim
  - Kliniken Maria Hilf GmbH - Krankenhaus St. Franziskus, Mönchengladbach
  - Medizinische Klinik und Poliklinik III - Universitätsklinik, München
  - Klinikum Nuernberg, Nuremberg
  - Pi.Tri-Studien GmbH, Offenburg
  - CaritasKlinikum Saarbrücken, Saarbrücken
  - Marienhospital, Stuttgart
  - Klinik für Innere Medizin I, Ulm
  - Medizinische Studiengesellschaft NORD-WEST GmbH - Praxis Aurich, Westerstede
  - Medizinische Studiengesellschaft NORD-WEST GmbH, Westerstede
- St. László Teaching Hospital, Budapest, Hungary
- Switzerland (30):
  - Kantonsspital Aarau, Aarau
  - Kantonsspital Baden, Baden
  - Universitätsspital Basel, Basel
  - St. Claraspital Basel, Basel
  - IOSI, Ospedale San Giovanni, Bellinzona
  - Klinik Engeried / Oncocare, Bern
  - Inselspital Bern, Bern
  - Spitalzentrum Biel, Biel
  - Spitalzentrum Oberwallis, Brig
  - Kantonsspital Graubünden, Chur
  - HFR-Hôpital cantonal, Fribourg
  - CCAC Fribourg, Fribourg
  - Hopitaux Universitaires de Geneve, Geneva
  - Clinique de Genolier, Genolier
  - CCAC Lausanne, Lausanne
  - Centre Hospitalier Universitaire Vaudois, Lausanne
  - Kantonsspital Liestal, Liestal
  - Kantonsspital Luzern, Lucerne
  - Clinica Luganese, Lugano
  - Onkologie Zentrum Spital Männedorf, Manno
  - Spital Thurgau, Münsterlingen
  - Hôpital de Pourtalès, Neuchâtel
  - Kantonsspital Olten, Olten
  - Kantonsspital St. Gallen, Sankt Gallen
  - Spital Limmattal, Schlieren
  - Hôpital du Valais Sion, Sion
  - Bürgerspital Solothurn - Onkologiezentrum, Solothurn
  - SpitalSTS AG Simmental-Thun-Saanenland, Thun
  - Kantonsspital Winterthur, Winterthur
  - Stadtspital Zürich Triemli, Zurich

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Screened (n=1040) PIK3CA-mutated (n=180) Randomized (n=113)
  Excluded (n=67):
  * Not meeting inclusion criteria (n=20)
  * Declined to participate (n=43)
  * Other reasons (n=4)
Period: Allocation
Arm/Group | Aspirin 100 mg | Placebo
Started | 75 | 38
Completed | 74 | 38
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0
Period: Follow-up
Arm/Group | Aspirin 100 mg | Placebo
Started | 74 | 38
Completed | 63 | 29
Not Completed | 11 | 9
Not completed — Death | 5 | 4
Not completed — Lost to Follow-up | 6 | 5

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS): The FAS is defined as all randomized patients who received at least one dose of aspirin/placebo excluding patients with major eligibility violations as defined in the statistical analysis plan (SAP). Following the intention-to-treat principle, patients in this population were analyzed according to the treatment they were randomized to.
Groups:
- Total: Total of all reporting groups
Arm/Group | Aspirin 100 mg | Placebo | Total
Number analyzed (Participants) | 74 | 38 | 112
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 31 | 19 | 50
  >=65 years | 43 | 19 | 62
Age, Continuous [Median (Full Range); unit: years] | 68 [29 to 79] | 65 [44 to 89] | 66 [29 to 89]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 18 | 48
  Male | 44 | 20 | 64
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: African | 2 | 0 | 2
  Ethnicity: Asian | 3 | 0 | 3
  Ethnicity: Caucasian | 67 | 38 | 105
  Ethnicity: Hispanic | 1 | 0 | 1
  Ethnicity: Other | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  Belgium | 4 | 1 | 5
  Hungary | 1 | 1 | 2
  Switzerland | 44 | 25 | 69
  Germany | 25 | 11 | 36

OUTCOME MEASURES:

1. Primary Outcome: Disease-free Survival (DFS)
Description: The primary endpoint of this trial is DFS, defined as time from surgery until one of the following events, whichever comes first:
  * recurrence
  * second cancer
  * death due to any reason Patients not experiencing an event will be censored at the date of the last available tumor assessment.
Time Frame: up to 7 years
Measure: Median (95% Confidence Interval); unit: years
Arm/Group | Aspirin 100 mg | Placebo
Number analyzed (Participants) | 74 | 38
years | NA [6.19 to NA] — Not reached | NA [5.77 to NA] — Not reached
Statistical Analysis 1: Comparison: Aspirin 100 mg vs Placebo; Test type: Superiority; p = 0.11, Log Rank
Statistical Analysis 2: Comparison: Aspirin 100 mg vs Placebo; Test type: Superiority; Hazard Ratio (HR) = 0.57, 90% CI 2-sided [0.27 to 1.22] — Unstratified
Statistical Analysis 3: Comparison: Aspirin 100 mg vs Placebo; Test type: Superiority; Hazard Ratio (HR) = 0.57, 90% CI 2-sided [0.22 to 1.46] — Stratified

2. Secondary Outcome: Time to Recurrence (TTR)
Description: TTR was calculated from surgery until recurrence or death due to colon cancer. Patients not experiencing an event or patients who died due to other reasons before experiencing an event were censored at the date of the last available tumor assessment.
Time Frame: up to 7 years
Measure: Median (95% Confidence Interval); unit: years
Arm/Group | Aspirin 100 mg | Placebo
Number analyzed (Participants) | 74 | 38
years | NA [NA to NA] — Not reached | NA [5.77 to NA] — Not reached
Statistical Analysis 1: Comparison: Aspirin 100 mg vs Placebo; Test type: Superiority; p = 0.089, Log Rank
Statistical Analysis 2: Comparison: Aspirin 100 mg vs Placebo; Test type: Superiority; Hazard Ratio (HR) = 0.49, 90% CI 2-sided [0.21 to 1.19] — Unstratified
Statistical Analysis 3: Comparison: Aspirin 100 mg vs Placebo; Test type: Superiority; Hazard Ratio (HR) = 0.56, 90% CI 2-sided [0.20 to 1.55] — Stratified

3. Secondary Outcome: Overall Survival (OS)
Description: OS was calculated from surgery until death from any cause. Patients not experiencing an event were censored at the last date they were known to be alive.
Time Frame: up to 7 years
Measure: Median (95% Confidence Interval); unit: years
Arm/Group | Aspirin 100 mg | Placebo
Number analyzed (Participants) | 74 | 38
years | NA [NA to NA] — Not reached | NA [5.77 to NA] — Not reached
Statistical Analysis 1: Comparison: Aspirin 100 mg vs Placebo; Test type: Superiority; p = 0.3, Log Rank
Statistical Analysis 2: Comparison: Aspirin 100 mg vs Placebo; Test type: Superiority; Hazard Ratio (HR) = 0.71, 90% CI 2-sided [0.23 to 2.13] — Unstratified
Statistical Analysis 3: Comparison: Aspirin 100 mg vs Placebo; Test type: Superiority; Hazard Ratio (HR) = 0.60, 90% CI 2-sided [0.15 to 2.43] — Stratified

4. Secondary Outcome: Cancer-specific Survival (CSS)
Description: CSS was calculated from surgery until death due to colon cancer, whether due to the original tumor or to a second primary same cancer. Patients who died due to other reasons were censored at the time of death. All other patients were censored at the last date they were known to be alive.
Time Frame: up to 7 years
Measure: Median (90% Confidence Interval); unit: years
Arm/Group | Aspirin 100 mg | Placebo
Number analyzed (Participants) | 74 | 38
years | NA [NA to NA] — Not reached | NA [NA to NA] — Not reached

5. Secondary Outcome: Adverse Events (AEs)
Time Frame: During treatment (median 22.1 months)
Measure: Count of Participants; unit: Participants
Arm/Group | Aspirin 100 mg | Placebo
Number analyzed (Participants) | 74 | 38
Participants
  Anemia | 0 | 1
  Colonic hemorrhage | 0 | 1
  Cranial fracture with intra cranial hemorrhage | 0 | 1
  Dizziness | 1 | 0

ADVERSE EVENTS:
Time Frame: Deaths were assessed for up to 7 years. Adverse Events were assessed for an median of 22.1 months
Arm/Group | Aspirin 100 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 5/74 | 4/38
Serious Adverse Events (participants affected / at risk) | 1/74 | 3/38
Other Adverse Events (participants affected / at risk) | 0/74 | 0/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aspirin 100 mg (N=74) | Placebo (N=38)
Intraductal proliferative breast lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Colonic hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Cranial fracture with intracranial hemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
small sample size

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
SAKK GENERAL TERMS AND CONDITIONS (SAKK GTC) FOR TRIAL SPECIFIC AGREEMENTS

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-11-11): https://cdn.clinicaltrials.gov/large-docs/82/NCT02467582/Prot_SAP_000.pdf